CLINICAL TRIAL: NCT04275882
Title: Evaluation of Retrospective Demographic, Clinical and Etiologic Data of Patients Presenting to Cardiology Clinic and / or Outpatient Clinics With Left Ventricular Hypertrophy Detected by Electrocardiography and/or Echocardiography: LVH-TR
Brief Title: Demographical and Clinical Profile of Patients With Left Ventricular Hypertrophy
Status: Completed | Type: Observational
Sponsor: Cardiovascular Academy Society, Turkey (Other)
Responsible Party: Principal Investigator, Mehdi Zoghi, prof.dr., Cardiovascular Academy Society, Turkey
Other Study IDs: LVH-TR
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-08

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Echocardiography; retrospective; electrocardiography; hypertension; cardiomyopathy
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension; Cardiomyopathies | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Electrocardiogram — There will be no new intervention performed for the patients.
  Other Names: Echocardiography

SUMMARY:
Left ventricular hypertrophy (LVH) is the most common result of the heart trying to pump blood against the high afterload, as in hypertension and aortic stenosis.Although hypertension is the most common cause of LVH, LVH can also be found in athletes and cardiomyopathies or in storage disorders such as amyloidosis. In addition, genetic diseases also play an important role in the pathogenesis of LVH. Fabry disease is another disease that should be considered in patients with left ventricular hypertrophy.Left ventricular hypertrophy is a common and potentially modifiable cardiovascular risk factor that is frequently overlooked in clinical practice.The benefit of combining ECG and echocardiography in the diagnosis of LVH has been demonstrated.Early diagnosis and treatment-related regression of LVH, reduces adverse cardiovascular events and improves survival.Therefore, the investigators planned to perform a retrospective, observational LVH-TR study in order to determine the etiologic causes of LVH, the symptoms presented by the patients, and the effects of patients' demographic characteristics on LVH.

DETAILED DESCRIPTION:
Left ventricular hypertrophy (LVH) is an abnormal increase in the mass of the left ventricular (LV) myocardium caused by a chronic increased workload in the heart.This is most common result of the heart trying to pump blood against the high afterload, as in hypertension and aortic stenosis.Although hypertension is the most common cause of LVH, LVH can also be found in athletes and cardiomyopathies or in storage disorders such as amyloidosis. In addition, genetic diseases also play an important role in the pathogenesis of LVH. Fabry's disease is an X-linked lysosomal storage disorder caused by mutations in the gene encoding galactosidase A. In a study in which 47 patients analyzed, the prevalence of Fabry disease was found to be 2.1% in patients with LVH.Since enzyme replacement therapy is important for Fabry patients, early and accurate diagnosis is very important.Amyloidosis is another disease that should be considered in patients with left ventricular hypertrophy.It should be considered especially in patients with preserved ejection fraction heart failure, in patients over 60 years of age, in men with ventricular hypertrophy, and in case of incompatibility between left ventricular thickness and QRS voltage. In the THAOS study, symptoms and signs of cardiac involvement were found in 42.1% of patients with TTR amyloidosis. In a study that included of 3287 patients, the prevalence of LVH was 14.9% in men and 9.1% in women.LVH increases cardiovascular mortality and morbidity, so the etiology of LVH is extremely important to determine the method of treatment of patients and improve survival.Data from the Framingham Heart Study show that the presence of LVH diagnosed by ECG, X-ray, or echocardiography is associated with a 3-fold increased risk for CV events and 5 to 9-fold increased risk for sudden cardiac death.A meta-analysis based on 10 studies with 27,000 patients showed that LVH was associated with an increased risk of supraventricular and ventricular arrhythmias.The incidence of supraventricular tachycardia was 11.1% in patients with LVH and 1.1% in patients without LVH. The incidence of ventricular arrhythmia (tachycardia and fibrillation) was 5.5% in patients with LVH and 1.2% in patients without LVH.Several studies have shown that the risk of atrial fibrillation increases with LVH.As shown in the Framingham Heart Study, patients with atrial fibrillation are 5 times more likely to have a stroke and the mortality rate has increased by 1.5-1.9.

LVH can be detected by electrocardiography (ECG), echocardiography (ECHO) or cardiac magnetic resonance imaging (CMRI). Each has its own advantages and disadvantages.Among these tests ECG is the cheapest and easiest to diagnose LVH. Its specificity is acceptably high, but its sensitivity is low.Although ECG is not sensitive and is not used to rule out LVH, it still has a role in the diagnosis and management of LVH. The best-known electrocardiographic criteria for the diagnosis of LVH are the Cornell product and the Sokolow-Lyon index. Another preferred test for evaluating LVH is echocardiography. ECHO is much more sensitive than ECG, and it can also detect other abnormalities such as left ventricular dysfunction and valve disease. In this test, the left ventricular end-diastolic diameter, posterior wall thickness and interventricular septum thickness can be measured, and in addition to these measurements the left ventricular mass index can be calculated from the patient's height and weight.The benefit of combining ECG and ECHO to identify LVH has been documented. Patients with LVH on both ECG and ECHO have a particularly high risk of heart failure and hospitalization, so this indicating the importance of combining different methods for LVH assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have undergone ECG / ECO within the last 6 months and have been found to meet LVH according to the specified criteria
* older than 18 years and younger than 90 years
* who signed the informed consent form

Exclusion Criteria:

* Cases without optimal electro or echocardiographic examination due to limited echogenicity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to cardiology clinics and / or outpatient clinics with left ventricular hypertrophy (LVH) detected by ECG and / or echocardiography will be included retrospectively.
Sampling Method: Probability Sample
Enrollment: 886 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | 6 months
  Demographic characteristics of patients with left ventricular hypertrophy (LVH) on ECG and / or echocardiography
Evaluation of etiologic data | 6 months
  Evaluation of etiologic data of patients with left ventricular hypertrophy (LVH) on ECG and / or Echocardiography

OTHER OUTCOMES:
Frequency of Fabry and Amyloidosis | 6 months
  Frequency of Fabry and Amyloidosis in outpatient and / or hospitalized patients with LVH

CONTACTS AND LOCATIONS:
Overall Officials: mehmet kış, dr, Principal Investigator — turkey
Locations (1):
- Yasemin, Kayseri, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided